CLINICAL TRIAL: NCT05478083
Title: A GnRH Agonist IN Pre-menopausal Women STudy to Treat Severe Polycystic Liver Disease
Acronym: AGAINST-PLD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-005949-16; 2020-005949-16 (EudraCT Number); 10140261910001 (Other Grant/Funding Number: ZonMw); U1111-1278-8976 (Registry Identifier: Universal Trial Number (UTN))
Record Dates: First submitted 2022-05-09; First posted 2022-07-28 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Polycystic Liver Disease; Autosomal Dominant Polycystic Kidney
MeSH Terms: conditions — Polycystic liver disease; Polycystic Kidney, Autosomal Dominant | interventions — Leuprolide

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial in which patients are randomized between either 1. Direct start with treatment or 2. Delayed start with treatment which will start after 18 months of standard care with the study medication
Who Masked: Outcomes Assessor
Masking Description: Patient blinding is not possible, since leuprorelin will induce menopause related complaints.
  Primary outcome is not reported to investigators until the study has finished. Outcome assessors are blinded for study subject and treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct start (Active Comparator): 36 months of treatment with study medication
  Interventions: Drug: Leuprorelin
- Delayed start (Other): First 18 months standard care, hereafter 18 months treatment with study medication
  Interventions: Drug: Leuprorelin

INTERVENTIONS:
Drug: Leuprorelin — Treatment consist of leuprorelin 3.75 mg once monthly for the first 3 months followed by 3-monthly injections of 11.25 mg. The direct start group will use leuprorelin for 36 months. The delayed start group will use standard of care in the first 18 months.

SUMMARY:
Multicenter trial on the effect of the GnRH analogue leuprorelin on the growth of total liver volume in pre-menopausal women with very severe polycystic liver disease who, despite available therapy, experience growth and are heading for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Diagnosis of polycystic liver disease defined as the presence of more than 10 liver cysts
* Age between 18 to 45 (inclusive) years;
* Very large liver for age, defined as the upper 10% of liver volumes in specific age categories (based on a retrospective polycystic liver disease registry, n=1.600 patients)

  * 18-30 yr; height adjusted TLV > 2.0 L/m
  * 30-35 yr; height adjusted TLV > 2.2 L/m
  * 35-40 yr; height adjusted TLV > 2.5 L/m
  * 40-45 years; height adjusted TLV > 3.0 L/m
* Availability of at least 1 historical MRI or CT scan made between 5 to 1 years before baseline visit of this study
* Ongoing liver growth, defined as an increase in absolute total liver volume between the historical MRI or CT scan and the MRI at screening of this trial
* Since somatostatin analogues are proven efficacious therapy for polycystic liver disease at this time it is required that:

  * patients use a somatostatin analogue and still have confirmed liver growth; OR
  * patient have a specific reason not to use this medication, .e.g. patient used a somatostatin analogue in the past, but had to stop it due to inefficacy or because he/she did not tolerate it, patient has a contra-indication for using somatostatin analogues, no availability of somatostatin analogues
* Voluntary written informed consent before performance of any study-related procedures not part of standard medical care, and able to read, comprehend, and respond to study questionnaires.

Exclusion Criteria:

Post-menopausal status or (vasomotor) symptoms indicating upcoming menopause

* Anti Mullerian Hormone (AMH) measurement at screening visit <0.03 ng/ml.
* Active desire to have children, pregnancy or breast-feeding
* Contra-indications for leuprorelin, such as history of cardiovascular disease, history of osteoporosis or osteoporosis determined by DEXA-scan at screening (T score ≤ - 2.5), or a known intolerance for leuprorelin
* Liver transplantation or liver surgery expected within 1.5 years, to the discretion of the study doctor
* Use of hormonal oral contra-conception containing estrogen and/or progesterone. In contrast, a hormone containing uterine device is not an exclusion criteria.
* Contra-indications for MRI assessments (such as implants) or not able or willing to undergo MRI scan for other reasons (e.g. claustrophobia, profound obesity)
* Kidney transplantation or chronic use of immunosuppressive agents (such as cyclosporine, mycophenolic acid, tacrolimus but not prednisolone) for other indications
* Severe hypertension, defined as a systolic blood pressure >160 mmHg and/or diastolic blood pressure > 100 mm Hg.
* Clinically significant, uncontrolled medical condition that, in the opinion of the investigator, would put the safety of the patient at risk through participation, or which would affect the efficacy of safety analysis if the condition exacerbated during the study, or that may significantly interfere with study compliance, such as, but not restricted to, recurrent cholangitis, recurrent ascites or hepato-venous outflow obstruction, (history of) depression
* Participation in other interventional studies at the same time.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female hormones, especially estrogen, seem to play a pivotal role in liver growth. More than 90% of patients is female and exogenous estrogen administration enhances liver growth and liver growth declines after menopause.
Enrollment: 36 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Liver growth | 36 months
  Liver volumes (in % per year) measured in the MRI at screening, 6 months, 18 months, 24 months and 36 months

SECONDARY OUTCOMES:
Polycystic liver disease related complaints | 36 months
  PLD related complaints assessed by the Polycystic liver disease-Questionnaire at baseline, 6 months, 18 months, 24 months and 36 months
Menopause related complaints | 36 months
  Menopause related complaints by using the validated MENQOL questionnaire at baseline, 6 months, 18 months, 24 months and 36 months
Patient reported mental health | 36 months
  Quality of life and as subset mental health will be measured by the validated RAND SF-36 questionnaires at baseline, 6 months, 18 months, 24 months and 36 months
Patient reported physical health | 36 months
  Quality of life and as subset physical health will be measured by the validated RAND SF-36 questionnaires at baseline, 6 months, 18 months, 24 months and 36 months
Kidney growth | 36 months
  Kidney volumes (in % per year) measured in the MRI at screening, 6 months, 18 months, 24 months and 36 months
Sex hormone levels | 36 months
  Anti Muller Hormone will be assessed at screening. Other Extensive laboratory includes estradiol, progesterone, AMH, FSH, LH levels at baseline, 6 months after start therapy and after 18 and 36 months.
Bone density | 36 months
  Bone density measured by a DEXA scan at screening, 18 months and 36 months.
Renal function | 36 months
  eGFR measurements and 24h urine analyisis (in ADPKD patients only) at baseline, 6 months, 18 months, 24 months and 36 months time
Bloodpressure | 36 months
  Manual blood pressure measurements in millimetres of mercury (measure 3 times with 2 minutes in between) at screening, baseline, 3 months, 6 months, 12 months, 18months, 21 months, 24 months, 30 months and 36 months .
Heart rate | 36 months
  Heart rate in beats per minute (measure 3 times with 2 minutes in between) measured at screening, baseline, 3 months, 6 months, 12 months, 18months, 21 months, 24 months, 30 months and 36 months .
Weight | 36 months
  Body weight in kilograms measured at screening, baseline, 3 months, 6 months, 12 months, 18months, 21 months, 24 months, 30 months and 36 months .
Upper-arm-circumference | 36 months
  Upper-arm-circumference in centimeters of the non-dominant arm measured at screening, baseline, 3 months, 6 months, 12 months, 18months, 21 months, 24 months, 30 months and 36 months.
Abdominal circumference | 36 months
  Abdominal circumference in centimeters (measured at the level of the umbilicus) measured at screening, baseline, 3 months, 6 months, 12 months, 18months, 21 months, 24 months, 30 months and 36 months .
  At screening, length will be collected to calculate Body Mass Index.
Length | 1 month
  At screening length in centimeters will be collected.
The number of participants experciencing a (serious) adverse events | 36 months
  During each physical or telephone contact, the adverse effects are queried and registered in accordance with national protocol
Symptoms of depression | 36 months
  Symptoms of depression measured by the validated BD-II questionnaires at baseline, 6 months, 18 months, 24 months and 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Groningen universitair medical center, Groningen

IPD SHARING:
Plan to Share IPD: No